CLINICAL TRIAL: NCT03133988
Title: An Expanded Access Program Providing Margetuximab in the Treatment of HER2+ Metastatic Breast Cancer in Single, Individually-approved Patients
Brief Title: Margetuximab Expanded Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: TerSera Therapeutics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MGAH22-EA
Record Dates: First submitted 2017-04-20; First posted 2017-04-28 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Carcinoma
MeSH Terms: interventions — margetuximab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: Margetuximab — anti-HER2 monoclonal antibody
  Other Names: MGAH22

SUMMARY:
The purpose of the Expanded Access program is to provide margetuximab to patients with pretreated HER2+ breast cancer for whom potential benefit justifies potential treatment risks.

DETAILED DESCRIPTION:
TerSera Therapeutics LLC (TerSera) will consider, on a case-by-case basis, requests by treating physicians to file a single patient investigational new drug application for expanded access to margetuximab and for TerSera to supply margetuximab for single patient use.

ELIGIBILITY:
Inclusion Criteria:

* TerSera may consider requests on a case-by-case basis from treating physicians for patients not otherwise eligible for margetuximab clinical studies.
* Treating physicians should consider approved therapies for a patient's disease, as well as ongoing clinical studies, before seeking expanded access use with an investigational agent.

Exclusion Criteria:

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult